CLINICAL TRIAL: NCT01334203
Title: A Phase 4, Randomized, Double-Blind, Placebo-Controlled, Parallel Study of Ranolazine in Subjects With Chronic Stable Angina and Coronary Artery Disease With a History of Type 2 Diabetes Mellitus
Brief Title: A Study on the Effects of Ranolazine on Exercise Duration in Subjects With Chronic Stable Angina and Coronary Artery Disease (CAD) With Type 2 Diabetes Mellitus (T2DM)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Jay Garg, MD, Director, Clinical Research, Gilead Sciences, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-259-0108
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Angina Pectoris; Coronary Artery Disease; Type 2 Diabetes Mellitus
Keywords: Chronic angina; Angina pectoris; Coronary artery disease; Type 2 Diabetes Mellitus; ETT
MeSH Terms: conditions — Angina Pectoris; Coronary Artery Disease; Diabetes Mellitus, Type 2 | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranolazine (Experimental)
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator)
  Interventions: Drug: Ranolazine

INTERVENTIONS:
Drug: Ranolazine — Subjects will be randomized to either ranolazine 500 mg twice daily up-titrated on Day 4 to 1000 mg administered orally twice a day or matching placebo for the 12 week treatment period.
  Subjects receiving diltiazem or verapamil as their concomitant antianginal medication will receive ranolazine 500 mg or placebo administered orally twice a day.
  Other Names: Ranexa

SUMMARY:
This study will evaluate the efficacy of ranolazine compared to placebo on duration of exercise assessed by exercise tolerance testing (ETT) at anticipated peak ranolazine plasma concentration after 12 weeks of treatment in subjects with chronic stable angina and coronary artery disease (CAD) who have a history of type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
This study will evaluate the efficacy of ranolazine compared to placebo on duration of exercise assessed by exercise tolerance testing (ETT) at anticipated peak ranolazine plasma concentration after 12 weeks of treatment in subjects with chronic stable angina and coronary artery disease (CAD) who have a history of type 2 diabetes mellitus (T2DM). This is a randomized, double-blind, placebo-controlled, parallel group study in subjects with chronic stable angina and CAD receiving a stable dose of a single concomitant antianginal medication who also have a history of T2DM; allowed antianginals will be a beta-blocker (atenolol or metoprolol) or a calcium-channel blocker.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Males and females aged 18 to 79 years
* Able to perform a Sheffield Modified Bruce Treadmill Exercise Protocol
* At least a 3-months history of chronic stable angina triggered by physical effort and relieved by rest and/or sublingual nitroglycerin
* Coronary artery disease documented by one or more of the following:

  * Angiographic evidence of ≥ 50% stenosis of one or more major coronary arteries
  * History of myocardial infarction (MI) documented by positive CK-MB enzymes, troponins, or ECG changes
  * Cardiac nuclear scan studies diagnostic of CAD, e.g., thallium scan or ECHO with stress or pharmacologic interventions (adenosine, dipyridamole, etc.)
* Stable treatment with one of the following antianginal medications for at least 4 weeks prior to Screening:

  * beta-blocker (atenolol up to 50 mg daily or metoprolol up to 100 mg daily)
  * dihydropyridine calcium-channel blocker (amlodipine up to 5 mg daily or nifedipine up to 30 mg daily)
  * non-dihydropyridine calcium-channel blocker (diltiazem 180 to 360 mg daily or verapamil 180 to 360 mg daily)
* Willingness to discontinue other antianginals and be treated with one of the allowed antianginal therapies
* Documented history of type 2 diabetes mellitus
* Females of childbearing potential must agree to utilize highly effective contraception methods from Screening throughout the duration of study treatment and for 14 days following the last dose of study drug.

Exclusion Criteria:

* Inability to exercise or having exercise limitation due to other co-morbidities that may interfere with ability to perform required ETT (e.g., morbid obesity, significant chronic lung disease, prior hospitalization for acute exacerbation of chronic lung disease or home oxygen use, chronic oral steroid therapy that can limit exercise capacity, osteoarthritis, peripheral artery disease, etc.)
* Any absolute contraindication to ETT
* Presence of electrocardiographic or other abnormalities that interfere with ECG interpretation or may cause a false positive stress test (e.g., ≥ 1 mm horizontal or down-sloping ST segment depression at rest in any standard ECG lead, Lown-Ganong-Levine syndrome, Wolff-Parkinson-White syndrome, left bundle branch block, left ventricular hypertrophy with repolarization abnormality, ventricular pacemaker, etc.)
* Decompensated heart failure
* Clinically significant valvular heart disease or congenital cardiac defects
* Acute coronary syndrome in the prior 2 months or coronary revascularization within the prior 6 months or planned coronary revascularization during the study period
* Stroke or transient ischemic attack within 6 months prior to Screening
* History of serious ventricular dysrhythmias or a history of life-threatening ventricular arrhythmia
* Atrial fibrillation
* QTc > 0.5 seconds
* Hypertrophic cardiomyopathy
* Uncontrolled hypertension (seated systolic blood pressure > 180 mm Hg or diastolic blood pressure > 110 mm Hg)
* Systolic blood pressure < 90 mm Hg
* Inability to discontinue current antianginal medications and remain on one allowed antianginal therapy
* Clinically significant hepatic impairment
* Creatinine clearance (CLCr) < 30 ml/min
* Prior treatment with ranolazine
* Participation in another investigational drug or device study within 1 month prior to Screening
* Females who are breastfeeding
* Positive serum pregnancy test
* Current treatment with potent inhibitors of CYP3A (e.g., ketoconazole, itraconazole, clarithromycin, nefazodone, nelfinavir, ritonavir, indinavir, and saquinavir)
* Current treatment with CYP3A and P glycoprotein (Pgp) inducers (e.g., rifampicin/rifampin, carbamazepine, St. John's wort)
* History of illicit drug use or alcohol abuse within one year of screening
* Any other conditions that, in the opinion of the investigator, are likely to prevent compliance with the study protocol or pose a safety concern if the subject participates in the study

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the change from baseline in exercise treadmill duration in the peak ETT at week 12 or last visit. | 12 weeks

SECONDARY OUTCOMES:
Time to onset of angina during peak ETT at week 12 or last visit | 12 weeks
Time to onset of 1 mm ST-segment depression during peak ETT at week 12 or last visit | 12 weeks
Change from baseline in exercise treadmill duration in the trough ETT at week 12 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jay Garg, MD, Study Director — Gilead Sciences